CLINICAL TRIAL: NCT07139639
Title: Evidence-Based Evaluation and New Drug Development of Classic Herb Pair (Chuanxiong Rhizoma and Salviae Miltiorrhizae) for Preventing Recurrence of Diabetic Lower Extremity Arterial Disease
Brief Title: Evidence-Based Evaluation of Classic Herb Pair (Chuanxiong Rhizoma and Salviae Miltiorrhizae) for Preventing Recurrence of Diabetic Lower Extremity Arterial Disease
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zheng Liu (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); Peking University Third Hospital (Other); Dongzhimen Hospital, Beijing (Other); Xuanwu Hospital, Beijing (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Zheng Liu, MD-PhD, Affiliated Hospital of Shandong University of Traditional Chinese Medicine
Organization: Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025-035-03-KY; 2024ZD0532600, 2024ZD0532603 (Other Grant/Funding Number: National Health Commission Science & Technology Development Research Center)
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Lower Extremity Arterial Disease
Keywords: Recurrence of ulcer; Diabetic Lower extremity arterial disease; Interventional Study; Prevention; Guanxinning Tablets; Salviae Miltiorrhizae; Chuanxiong Rhizoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Background Therapy Strict dietary control
  Standardized medication Administered according to glycemic, lipid, and blood pressure treatment guidelines
  Individualized antithrombotic regimen:
  * First-line: Aspirin 100mg/d
  * Alternative: Clopidogrel 75mg/d or other antithrombotic agents if aspirin allergy Note: Specific interventions adjusted based on actual clinical conditions Experimental Arm Background therapy + Guanxinning Tablets
  Interventions: Drug: Guanxinning Tablets
- Placebo Arm (Placebo Comparator): ackground Therapy Strict dietary control
  Standardized medication Administered according to glycemic, lipid, and blood pressure treatment guidelines
  Individualized antithrombotic regimen:
  * First-line: Aspirin 100mg/d
  * Alternative: Clopidogrel 75mg/d or other antithrombotic agents if aspirin allergy Note: Specific interventions adjusted based on actual clinical conditions Placebo Arm Background therapy + Matching Placebo for Guanxinning Tablets
  Interventions: Drug: Matching Placebo for Guanxinning

INTERVENTIONS:
Drug: Guanxinning Tablets — Guanxinning Tablets
  * Manufacturer: Zhengda Qingchunbao Pharmaceutical Co., Ltd.
  * NMPA Approval No. Z20150028
  * Administration: 4 tablets orally, three times daily for 6 months
  Arms: Experimental Arm
Drug: Matching Placebo for Guanxinning — Matching Placebo for Guanxinning Tablets
  * Manufacturer: Zhengda Qingchunbao Pharmaceutical Co., Ltd.
  * Drug Product Certificate of Analysis Approval No.YF-R-C037A-2024104-A
  * Administration: 4 tablets orally, three times daily for 6 months
  Arms: Placebo Arm

SUMMARY:
Taking the approach of promoting qi circulation and activating blood as the entry point, this study targets lower extremity arterial disease（LEAD） patients with TCM syndrome pattern of blood stasis due to qi stagnation. Using Guanxinning Tablets (a herbal formula with qi-moving and blood-activating properties) as the investigational medication, we will conduct a multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of the classic herb pair (Chuanxiong Rhizoma-Salviae Miltiorrhizae) in preventing LEAD ulcer recurrence. This research aims to accumulate evidence-based medical data supporting new drug development.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 80 years old (inclusive)
2. Diagnosis: Confirmed type 1 or type 2 diabetes mellitus
3. Meeting diagnostic criteria for diabetic lower extremity arterial disease (DLEAD)
4. TCM Syndrome: Qualified for Qi Stagnation and Blood Stasis syndrome pattern
5. Glycemic Control:

   * HbA1c ≤9% or Fasting plasma glucose ≤10 mmol/L
6. Ulcer History:

   * Documented history of diabetic lower extremity arterial disease (DLEAD)-related ulcers, with confirmed healing (wound re-epithelialization without signs of redness, purulent discharge, or infection) 2-8 weeks prior to enrollment.
7. Consent: Voluntarily signed informed consent form

Exclusion Criteria:

* (1) Ulcer Etiology Exclusion:
* Pure pressure ulcers
* Pure neuropathic ulcers
* Immune-mediated ulcers (e.g., vasculitic ulcers caused by lupus, Behcet's disease, rheumatoid arthritis) (2) Recent Cardiovascular Events:
* Acute coronary syndrome within 3 months
* Hemorrhagic stroke within 3 months (3) Organ Dysfunction:
* Severe hepatic impairment (AST or ALT >1.5×ULN)
* Chronic kidney disease stage 4-5 (eGFR <30 mL/min/1.73m²) (4) Recent Major Bleeding:
* Gastrointestinal hemorrhage within 1 month (5) Concurrent TCM Therapy:
* Use of blood-activating/stasis-resolving TCM preparations for DLEAD within 1 week (6) Herbal Contraindication:
* Concurrent or planned use of *Veratrum*-containing preparations (7) Malignancy:
* Active cancer progression (8) Reproductive Status:
* Pregnant or lactating women (9) Allergy History:
* Known hypersensitivity to *Ligusticum chuanxiong* or *Salvia miltiorrhiza* (10) Cognitive/Language Barriers:
* Psychiatric disorders
* Intellectual/language impairment affecting scale completion
* Unwillingness to cooperate (11) Life Expectancy:
* <1 year (12) Clinical Trial Participation:
* Enrollment in other drug trials within 1 month (13) Investigator's Discretion:
* Other conditions deemed unsuitable for participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Ulcer Recurrence Rate | Measured at 6 months post-intervention
  Ulcer Recurrence Rate = (Number of Subjects with Recurrent Ulcers / Total Subjects) × 100%

SECONDARY OUTCOMES:
Ulcer Recurrence Rate | Ulcer recurrence rates at 3, 9, and 12 months post-intervention
  Ulcer Recurrence Rate = (Number of Subjects with Recurrent Ulcers / Total Subjects) × 100%
Calculation of ulcer recurrence episodes | Assessed at 6 months post-intervention
  Recurrence is counted based on the timing of occurrence. Ulcers appearing concurrently at distinct anatomical sites are counted as one episode; those occurring at different time points are counted as multiple episodes.
Ankle-Brachial Index | 6 and 12 months after intervention
TCM Syndrome Score | at 3 and 6 months post-intervention
  TCM Syndrome Scoring Scale Description
  This scale quantifies six core manifestations of Qi Stagnation and Blood Stasis Syndrome in diabetic lower extremity arterial disease, using a four-tier scoring system (0/2/4/6 points):
  Limb coldness: Asymptomatic (0 pts); Occasional, self-relieved (2 pts); Persistent, relieved by warmth (4 pts); Persistent, unrelieved by warmth (6 pts)
  Limb pain: None (0 pts); Mild (2 pts); Moderate (4 pts); Severe (sleep-disturbing) (6 pts)
  Chest/abdominal distension: Absent (0 pts); Occasional mild (2 pts); Frequent moderate (4 pts); Frequent severe (6 pts)
  Skin temperature: Normal (0 pts); Slightly decreased (2 pts); Significantly decreased (4 pts); Cold (6 pts)
  Intermittent claudication: Absent (0 pts); Distance >500 meters (2 pts); 200-500 meters (4 pts); ≤200 meters (6 pts)
  Foot coloration: Normal (0 pts); Dark red (2 pts); Pale/purplish-dark (4 pts); Cyanosis/ecchymosis (6 pts)
Major Adverse Cardiovascular and Cerebrovascular Events (MACCE)、All-Cause Mortality | 3, 6, 9, and 12 months after intervention

IPD SHARING:
Plan to Share IPD: Yes